CLINICAL TRIAL: NCT02057536
Title: Pilot Study for the Effect of Exercise Intervention in Breast Cancer Patients With Arthralgias Receiving Aromatase Inhibitors
Brief Title: The Effect of an Exercise Program in Breast Cancer Patients With Joint Pain While Taking Aromatase Inhibitors.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCC# 34006
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Women With ER Positive Breast Cancer Taking (AI) w Joint Discomfort and Stiffness
Keywords: estrogen receptor positive, aromatase inhibitors, exercise,
MeSH Terms: conditions — Motor Activity | interventions — Observation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): 8 week directed exercise program
  Interventions: Other: Arm A Directed exercise program
- Arm B (Active Comparator): No directed exercise other than patients normal level of activity
  Interventions: Other: Observation

INTERVENTIONS:
Other: Arm A Directed exercise program
  Arms: Arm A
Other: Observation
  Arms: Arm B

SUMMARY:
The objective of this study is to determine if patients taking aromatase inhibitors (AI), who are experiencing joint discomfort and stiffness, would have reduction in this discomfort and stiffness by participating in a directed exercise program. The overarching objective is to improve patient compliance with the medication and ultimately clinical outcome.

In this pilot study, we will utilize a scientific approach for proof of concept employing both objective (inflammatory cytokine profiles and Physical Therapy (PT) measurements) and subjective (patient perception) methods to support an evidence based clinical plan. Patients will be divided into two cohorts. Group A will receive AI therapy with a directed exercise program. Group B will receive AI therapy without a directed exercise program. Data will be collected when both cohorts of patients enroll in the study, at the end of PT for Group A and, at the end of 8 weeks for Group B. At these time points, both groups will undergo a PT evaluation; have blood drawn for cytokine profiles; answer questions on an iPad that includes: the Pain Disability Index, the PHQ-4 (Psycological Health Questionaire depression scale, and pain level scale.

ELIGIBILITY:
Inclusion Criteria:

* 1. Women over age 40 with histological evidence of hormone receptor positive breast cancer.

  2. Post- menopausal 3. Adjuvant AI therapy. 4. Significant joint discomfort/stiffness when attempting activities of daily living which began or significantly increased after initiation of AI therapy.

  5. Currently not in an active directed exercise program (>60 minutes 2x/wk)

Exclusion Criteria:

1. Preexisting RA or fibromyalgia. 2. Systemic metastasis 3. ECOG performance status of greater than 2.

-

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Pain Disability Index | 8 weeks
  directed exercise program will improve patient response to the pain disability index survey.

SECONDARY OUTCOMES:
Plasma levels of inflammatory markers. | 8 weeks
  compare levels pre and post levels of markers in patient's plasma by an ELISA panel from patients in both arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Christiana Care/Helen F. Graham Cancer Center, Newark, Delaware, United States